CLINICAL TRIAL: NCT07405424
Title: Spiritual Care to Optimize Relationships and Experience in Adults With Acute Leukemia (SCORE Trial)
Brief Title: Spiritual Care Intervention in Adult Patients Diagnosed With Acute Leukemia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB25-0210
Record Dates: First submitted 2025-12-15; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spiritual Intervention Arm (Experimental): Participants receive a study specific spiritual care intervention.
  Interventions: Behavioral: SCORE Intervention
- No Intervention Arm (No Intervention)

INTERVENTIONS:
Behavioral: SCORE Intervention — Participants assigned to this arm will receive regularly scheduled visits from the study spiritual care team during their hospital admission (four times within 14 days).
  Arms: Spiritual Intervention Arm

SUMMARY:
This study is being done to determine if it is possible to incorporate spiritual care sessions as part of the care plan for patients hospitalized for leukemia treatment. In this study, participants will be randomly assigned to either no intervention (standard, real world inpatient spiritual care) or to receive study-specific guided spiritual sessions.

ELIGIBILITY:
Inclusion criteria

* Adults (18 years or older)
* Diagnosis of Acute Leukemia (AML or ALL) undergoing inpatient initial therapy
* Ability to read, understand, and speak the English language
* Ability to understand and the willingness to sign a written informed consent document

Exclusion criteria

* Unable to comply with spiritual care intervention
* Relapsed or refractory acute leukemia
* Cognitive deficits that limit participation and survey questionnaire completion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-06-20 (Estimated); Primary Completion 2028-06-16 (Estimated); Study Completion 2028-06-16 (Estimated)

PRIMARY OUTCOMES:
Is it feasible to enroll patients to a spiritual intervention study? | End of study (approximately 2 years)
  Study will compare the number of potential participants to those that enroll and complete 3 out of 4 study intervention sessions.
Will patients accept using the study specific spiritual intervention? | End of study (approximately 2 years)
  This will be measured on using the Lothian Chaplaincy Patient Reported Outcome Measure (PROM) questionnaire. This measures patient feelings related to spiritual care using rating from not at all to all of the time.

SECONDARY OUTCOMES:
Improvement on Patient Reported Spiritual Wellness | End of study (approximately 2 years)
  This will be measured by improvement (higher scores) reported by participants on the Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being 12 Item Scale (FACIT-sp12) questionnaire.
Improvement on Patient Reported Quality of Life | End of study (approximately 2 years)
  This will be measured by improvement (higher scores) reported by participants on the Functional Assessment of Cancer Therapy - Leukemia (FACT-Leu) questionnaire.
Improvement on Patient Reported Mood | End of study (approximately 2 years)
  This will be measured by improvement (lower scores) reported by participants on the Hospital Anxiety and Depression Scale (HADS) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Stock, Principal Investigator — University of Chicago
Locations (1):
- UChicago Medicine Comprehensive Cancer Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No